CLINICAL TRIAL: NCT04892004
Title: Does Symptom Recognition Improve Self-care in Patients With Heart Failure. A Growth Latent Model
Brief Title: Symptom Recognition Improves Self-care in Patients With Heart Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Joana Sousa, PhD, Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SympRecgHF
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure; Symptoms and Signs
Keywords: Heart failure; Self-care behaviors; Symptom recognition; Nurse-led program
MeSH Terms: conditions — Heart Failure; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard information defined as the standard care, unplanned, provided for Heart Failure patients and not personalized.
- Interventional group (Experimental): A nurse provides the intervention with expertise in Heart Failure and addresses reinforcements on: a) an explanation on signs and symptoms of Heart Failure and how to recognise them; b) importance on daily fluid management, by planning 1.5-2 litres of liquids per day (e.g., soup, milk, coffee, water, tea and yoghurts); and c) when doctors or nurses should be contacted (when symptoms escalation or a weight gain of 2 kg in three days or 5 kg in a week were detected).
  Interventions: Behavioral: Symptom recognition

INTERVENTIONS:
Behavioral: Symptom recognition — The patient receives a leaflet, which includes information about HF, primary symptoms, awareness of its detection and the fluid management plan. It also receives a weight diary, which helps him/her recall weight fluctuation and contact the nurse or doctor to call for help in a previous stage and avoid hospitalisation. Patients have to explain what they understand by HF, on follow-ups contacts, which are the main symptoms, if they are experiencing any of them and which difficulties managing fluid restriction and weight control. The leading investigator validates the information and teaches back contents if required.
  Arms: Interventional group

SUMMARY:
Describe a behaviour intervention to analyse self-care engagement in heart failure patients. Allocate patients with heart failure into 2 arms study: a control group and an intervention group.

DETAILED DESCRIPTION:
According to medical record at admission, a pilot study was described and included 63 patients in New York Heart Association (NYHA) functional class II-III. Patients were recruited in a hospital setting after discharge from a heart failure unit.

Patients were allocated into a control group (n=33) and an intervention group (n=30) through the computerised random allocation generator at http://random.org.

The pilot study was performed during three months per patient, with four moments of assessment (baseline, first-week follow-up, first-month follow-up, third-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* adults aged >18 years old, with diagnosed HF and with no cognitive disability associated.

Exclusion Criteria:

* patients placed on the heart transplant waiting list and patients in class IV NYHA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Symptom recognition | up to 3 months
  Awareness by a person of the body changes and how they can affect him/her
Self-care behaviors | up to 3 months
  Analyze if self-care behaviors are improved
Emergency and Hospital admissions | up to 3 months
  Report if patients with Heart Failure are admitted into hospital or emergency room

REFERENCES:
- [Derived] Pereira Sousa J, Neves H, Pais-Vieira M. Does Symptom Recognition Improve Self-Care in Patients with Heart Failure? A Pilot Study Randomised Controlled Trial. Nurs Rep. 2021 Jun 1;11(2):418-429. doi: 10.3390/nursrep11020040. PMID 34968218